CLINICAL TRIAL: NCT05533346
Title: Long-term Effects of WISE Program Improving Frailty Status and Quality of Life for Adolescents With Congenital Heart Disease
Brief Title: Long-term Effects of WISE Program Improving Frailty Status and Quality of Life for Adolescents With CHD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on our previous investigations, we've decided to construct a scale first.
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202112099RINA-202200361B0
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2022-09

CONDITIONS: Frailty
Keywords: CHD, adolescents, quality of life, walking
MeSH Terms: conditions — Frailty | interventions — SOSTDC1 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental - with WISE (Experimental): The experimental group will provide walking health education leaflets and exercise measurement wristbands for exercise monitoring, and will be given the intervention of the WISE program: three times a week, each time walking for at least 30 minutes, with a pace between 100-130 steps/ minutes, and then increase the number or time weekly according to personal ability.
  Interventions: Behavioral: with WISE (Walking Instruction based on Self-Efficacy)
- Control - without WISE (Active Comparator): The procedure of the control group will be the same as that of the experimental group, providing walking and health education leaflets and exercise measurement wristbands for exercise monitoring, but no intervention in the WISE program.
  Interventions: Behavioral: without WISE (Walking Instruction based on Self-Efficacy)

INTERVENTIONS:
Behavioral: with WISE (Walking Instruction based on Self-Efficacy) — Will be provided with walking health education leaflets and exercise measurement wristbands for exercise monitoring. Only the experimental group will be additionally given the interventional treatment of the WISE program: walk three times a week for at least 30 minutes each time, with a pace between 100-130 steps/min, and then increase the number or time weekly according to your personal ability, and remind you if the monitoring heart rate is higher than 170 times/min or the blood oxygen concentration is lower than 95%, and if the body feels any discomfort, it is necessary to stop taking a rest, and an educational strategy for improving self-efficacy of walking for 12 weeks is also provided.
  Arms: Experimental - with WISE
Behavioral: without WISE (Walking Instruction based on Self-Efficacy) — The procedure of the control group was the same as that of the experimental group, both of which will be provided with walking health education leaflets and exercise measurement wristbands for exercise monitoring.
  Arms: Control - without WISE

SUMMARY:
Most children with congenital heart disease (CHD) are expected to survive until adulthood. In addition to physical limitations, the growing adolescents with CHD are also challenged at the psychosocial domains. Previous studies have investigated the frailty of elderly, but the research on the intervention to the frailty of adolescents with CHD has been limited. The aims of this study will apply the Walking Instruction based on Self-Efficacy (WISE) program to examine the long-term effects of improving frailty state and quality of life for adolescents with CHD.

DETAILED DESCRIPTION:
This proposal will conduct a three-year series of studies. In the first year, a cross-sectional survey will be used to evaluate the applicability of the Fried frailty index to adolescents with CHD, and to examine the correlation between frailty index and quality of life in adolescent patients. In the second year, investigators will conduct individual in-depth interviews with selected pre-frailty/frailty adolescent participants and their main caregivers to gain insights into their views, connotations and support needs for frailty, which will serve as the basis for the design of the next interventional study. In the third year, the WISE program will be developed to provide 12-week walking self-efficacy improvement education strategies and exercise bracelets with heart rate monitoring. The recruited pre-frailty/frailty adolescent participants will be randomly assigned to experimental and control groups respectively in the pretest-posttest control group design. The changes in frailty state and quality of life for the two groups will be evaluated at 6, 12 and 24 weeks. The results of this study can provide frailty evaluation indicators for adolescents with CHD, timely detect the pre-frailty stage, and provide an important reference for the prevention of frailty intervention for adolescents with CHD as early as possible.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 12-18 years old.
2. Congenital heart disease diagnosed by a doctor before the age of 2.
3. The American New York Heart Association (NYHA) classifies the cardiac function as I-III grades.
4. Adolescents and their parents or guardians can communicate in Mandarin and Taiwanese and have normal cognitive abilities.
5. Those who are willing to cooperate with the research and complete the consent form.

Exclusion Criteria:

1. Received a heart transplant within one year.
2. Have undergone open-heart surgery within six months.
3. The New York Heart Association (NYHA) classifies the cardiac function as class IV.
4. Combined with other congenital diseases.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Frailty Status | change from baseline to post-intervention at 6-week follow-up
  The frailty phenotype and measurement method proposed by Fried et al. (2001) were modified to be suitable for use by adolescents. The five aspects of the assessment included decreased muscle strength, slow walking, thin body composition, self-reported fatigue and Decreased physical activity.
Frailty Status | change from baseline to post-intervention at 12-week follow-up
  The frailty phenotype and measurement method proposed by Fried et al. (2001) were modified to be suitable for use by adolescents. The five aspects of the assessment included decreased muscle strength, slow walking, thin body composition, self-reported fatigue and Decreased physical activity.
Frailty Status | change from baseline to post-intervention at 24-week follow-up
  The frailty phenotype and measurement method proposed by Fried et al. (2001) were modified to be suitable for use by adolescents. The five aspects of the assessment included decreased muscle strength, slow walking, thin body composition, self-reported fatigue and Decreased physical activity.

SECONDARY OUTCOMES:
Quality of life for adolescents with congenital heart disease | change from baseline to post-intervention at 6-week follow-up
  Quality of life scale for adolescents with congenital heart disease (PedsQLTM 3.0 Cardiac Module) will be used to measure participant's quality of life. This scale is divided into five aspects for measurement, including disease status, physical appearance, treatment anxiety, cognitive status and communication ability assessment. Those who take heart disease medicines must answer a total of 27 questions; those who do not take heart disease medicines have 22 questions, and each question has five options. 1 point for "yes", 2 points for "sometimes", 3 points for "often", and 4 points for "almost always". The lower the score, the better the quality of life.
Quality of life for adolescents with congenital heart disease | change from baseline to post-intervention at 12-week follow-up
  Quality of life scale for adolescents with congenital heart disease (PedsQLTM 3.0 Cardiac Module) will be used to measure participant's quality of life. This scale is divided into five aspects for measurement, including disease status, physical appearance, treatment anxiety, cognitive status and communication ability assessment. Those who take heart disease medicines must answer a total of 27 questions; those who do not take heart disease medicines have 22 questions, and each question has five options. 1 point for "yes", 2 points for "sometimes", 3 points for "often", and 4 points for "almost always". The lower the score, the better the quality of life.
Quality of life for adolescents with congenital heart disease | change from baseline to post-intervention at 24 week follow-up
  Quality of life scale for adolescents with congenital heart disease (PedsQLTM 3.0 Cardiac Module) will be used to measure participant's quality of life. This scale is divided into five aspects for measurement, including disease status, physical appearance, treatment anxiety, cognitive status and communication ability assessment. Those who take heart disease medicines must answer a total of 27 questions; those who do not take heart disease medicines have 22 questions, and each question has five options. 1 point for "yes", 2 points for "sometimes", 3 points for "often", and 4 points for "almost always". The lower the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No